CLINICAL TRIAL: NCT06367244
Title: Exercise and Wellness Behaviour Change for Solid Organ Transplant: A Hybrid Effectiveness-Implementation Trial of the Transplant Wellness Program
Brief Title: Transplant Wellness Program
Acronym: TWP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Stefan Mustata, Clinical Associate Professor, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TWP2023
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Transplantation
Keywords: Organ transplantation; Exercise; Prehabilitation; Health promotion; Behavior change; Rehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Liver Extracts

STUDY DESIGN:
Intervention Model Description: The TWP is a parallel study design with two arms. Participants are assigned to either the kidney or liver arm depending on the organ transplant they are listed or in evaluation for. Each arm will have a pre- or post- transplant group. Participants will be assigned to group depending on length of time between study enrollment and transplant surgery. Those with more than 12-weeks until surgery will complete the TWP pre-transplant and those with less than 12-weeks will complete the TWP post-transplant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kidney transplant arm (Experimental): Kidney transplant patients will be assigned to the kidney transplant arm and receive the standard 12-week exercise intervention in the TWP. Specific to the kidney arm will be certain patient reported outcomes (PROs). The Kidney Disease Quality of Life-36 (KDQOL-36) is a short form survey widely used to measure patient-reported QOL in patients on dialysis and is a validated tool in kidney transplant patients. Participants in the kidney arm will also receive disease-specific exercise and wellness materials to support their behaviour change.
  Interventions: Behavioral: Transplant Wellness Program - Kidney and Liver
- Liver transplant arm (Experimental): Liver transplant patients will be assigned to the liver transplant arm and receive the standard 12-week exercise intervention in the TWP. Specific to the liver arm will be certain PROs and functional fitness measures. The Chronic Liver Disease Questionnaire (CLQD) measures health-related QOL in patients with advanced liver disease and has been previously used in patients awaiting transplant. Liver arm participants will also complete the Liver frailty index, which requires a timed 5 sit-to-stands in addition to the other measures collected for the Fried Frailty Index. Participants in this arm will receive liver-specific exercise and wellness materials to support their behaviour change.
  Interventions: Behavioral: Transplant Wellness Program - Kidney and Liver

INTERVENTIONS:
Behavioral: Transplant Wellness Program - Kidney and Liver — The exercise prescription for the intervention will be multimodal, , will follow current chronic disease exercise guidelines, and will be tailored to meet the unique needs of each participant. . All participants will receive two 30-45-minute individual session with a CEP during their first week and two additional sessions during the second week if needed. The individual sessions will be followed by group sessions. Each participant will get a total of 24 individual and group sessions combined. These sessions can be conducted either in-person or online, based on participant preference and TWP logistics. For aerobic-based activities, a moderate rate of perceived exertion of 4-6 on a scale of 0-10 will be used. Resistance exercise will begin with functional movements and bodyweight exercises targeting major muscle groups with modifications for beginners and exercise progressions when deemed. Balance and flexibility training activities will also be included.

SUMMARY:
Wellness is defined as the active pursuit of activities, choices and lifestyles that lead to a state of overall health. Prehabilitation, or using rehabilitation in the period before surgery, can improve the pre, during, and post operative experience for the patient. Although exercise as prehabilitation has been well established in organ transplant, the investigators believe a multiphase approach will help to better serve patients and support patient wellness in the long-term. Supporting wellness behaviour change, such as exercise, stress reduction, and sleep, is associated with improved quality of life (QoL), mood, and improvements in well-being. Including behaviour change support in an exercise program can help support transplant patients in long-term positive lifestyle changes. The Transplant Wellness Program (TWP) is an exercise behaviour change program that includes additional wellness components such as nutrition, stress reduction, and sleep programs to support overall health and QoL of transplant patients. Specifically, the TWP will implement physical activity and behaviour change support for patients pre- and post-transplant surgery, addressing functional (frailty, indices of fitness, physical activity levels) and mental (anxiety, stress) outcomes to improve overall QoL. The TWP includes a 12-week exercise program that is delivered either pre-transplant or post-transplant, depending on length of time from study enrollment to transplant surgery. In addition to the exercise intervention, the TWP includes maintenance resources (access to group exercise classes, wellness webinars, group wellness coaching etc.), and wellness behaviour change support. The goal of the TWP is to improve outcomes of participants throughout their transplant journey, as well as reduce health services use. Collected outcomes will include program reach, effectiveness measures such as changes in physical fitness, adoption by healthcare practitioners, implementation of the program, and maintenance. In addition, will also collect health care use measures as the investigators believe the TWP will result in the reduction of several health care use outcomes, such as the number of hospital admissions (including intensive care unit admissions), length of hospital stays and emergency room utilization.

DETAILED DESCRIPTION:
Background and Rationale:

Wellness is defined as the active pursuit of activities, choices and lifestyles that lead to a state of holistic health. Prehabilitation, or using rehabilitation in the period before surgery, can help to optimize the surgical candidate and can improve the pre, peri and post operative experience for the patient. Although exercise as prehabilitation has been well established in solid organ transplant, the investigators believe a multiphasic approach will help to better serve patients and establish further health behavior change to support patient wellness in the long-term. Supporting wellness behaviour change, including using tenets from health coaching and patient-directed motivational counselling is associated with improved QOL, mood, and lowered perceived stress, as well as improvements in functional well-being. Incorporating behaviour change support in a multiphasic exercise prehabilitation program will support transplant patients in making positive lifestyle behaviour changes. Wellness programs need to be personalized and include behaviour change support to maintain motivation, provide feedback, and modify the program content as needed.

Research Question and Objectives: The Transplant Wellness Program (TWP) will target lifestyle behaviour change to enhance wellness, with a focus on improving exercise behaviour change. Specifically, the TWP will implement physical activity and behaviour change support for patients pre- and post-transplant surgery, addressing functional (frailty, indices of fitness, physical activity levels) and mental (anxiety, stress) outcomes to improve overall QOL. The goal of the TWP is to improve outcomes of participants throughout their transplant journey, as well as reduce health services utilization. In addition, the investigators believe the TWP will result in the reduction of several health care utilization outcomes, including the number of hospital admissions (including intensive care unit admissions), length of hospital stays and emergency room utilization. Finally, the TWP will also work in conjunction with additional resources across wellness, including nutrition services, stress reduction, and sleep programs, to support an integration of lifestyle modifiable behaviours that support enhanced well-being and quality of life.

Methods: The transplant wellness program (TWP) is intended to enhance wellness across the transplant trajectory. Introducing exercise and wellness behaviour change to support physical and psychosocial well-being before and after transplant surgery, the TWP will work closely with participants to tailor programming to meet their needs. The TWP specifically includes the Exercise Intervention (EI), which is a 12-week exercise program. EI is delivered either pre-transplant (EI-Pre-Transplant) or after transplant (EI-Post-Transplant) if patients are unable to participate before transplant. In addition to the exercise intervention, the TWP includes maintenance resources (access to group exercise classes, wellness webinars, group wellness coaching etc.), and wellness behaviour change support. The exercise intervention will be multiphasic (pre-transplant and post-transplant) and include wellness behavior change support. Implementation outcomes will be evaluated using the reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) framework.

To gain a better understanding of program implementation and to improve the quality of the program, participants will be requested to share their feedback upon completion of the exercise intervention through participant experience surveys and semi-structured interviews. Effectiveness outcomes include functional fitness outcomes (frailty and musculoskeletal function measures) and patient-reported outcomes (PROs). The PROs include QOL (using generic and disease specific measures), physical activity levels, sleep habits, nutrition, and mental health (anxiety and depression). Health economic evaluations will be performed to determine the cost-utility of implementing transplant wellness into the care pathway. Chart reviews will be done to collect information regarding outpatient and inpatient health care encounters, medication use, emergency visits, hospital admissions, length of hospital stays, intensive care unit admissions (length of stay and days intubated), patient and graft survival.

Procedures:

Study participants will complete functional fitness assessments across the TWP, including (i) at pre-intervention or intake; (ii) post-12-week exercise intervention (EI); and (iii) after surgery (12 weeks post). Follow-up assessments will occur at 6 months and 1-year post-EI intake. Participants will complete a wellness behaviour change support session before the12-week EI. The EI can be done before or after the transplant surgery. The functional fitness assessments and the wellness behaviour support session will take approximately 30 minutes each and can be done in-person or online based on logistics and participant preference. The functional fitness assessment will include: height and weight measurements, aerobic fitness test, muscular endurance test, and the standing balance test. The Patient Reported Outcome (PRO) questionnaires will be repeated at the same time points as functional fitness assessments and then annually for 5 years. Questionnaires will be done online (REDCap). The investigators will review the participants medical chart and collect medical history at the same time points.PRO questionnaires will take approximately 20 minutes to complete and be done online. These will be completed to assess: QOL, physical activity levels, diet, sleep habits, nutrition and mental health. Participants will be requested to share their feedback upon completion of the EI through participant experience surveys and semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* In evaluation or listed (active or temporarily inactive) on the transplant waiting list (kidney or liver) - status 0, 1, or 2
* Able to provide written informed consent and understand study information in English
* Approval to exercise from Canadian Society for Exercise Physiology - Clinical Exercise Physiologist (CSEP-CEP)
* Have access to an internet connected device

Exclusion Criteria:

* Not cleared for participation in the TWP by attending physician
* Unable to provide informed consent
* Clinical condition that makes the intervention unsafe or infeasible (e.g., unable to follow instruction due to refractory encephalopathy)
* Unsafe environment for virtual participation
* Recent variceal bleeding and cannot tolerate prophylaxis with non-selective beta blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2033-11 (Estimated); Study Completion 2033-11 (Estimated)

PRIMARY OUTCOMES:
Self-reported exercise | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 6-months post-intake, 1-, 2-, 3-, 4-, and 5- years post-intake.
  Change in self-reported exercise as assessed using the modified Godin Leisure Time Exercise Questionnaire (m-GLTEQ). Participants recall their typical weekly strenuous, moderate, and mild exercise. Each type of exercise is given a score and multiplied by the number of days per week the activity is performed. The sum of the items is then interpreted as either active (>24 points), moderately active (14-23 points), or insufficiently active/sedentary (<14 points).
Generic self-reported quality of life | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 6-months post-intake, 1-, 2-, 3-, 4-, and 5- years post-intake.
  Self-reported quality of life (QoL) is assessed by EuroQol- 5 Dimensions 5 Level (EQ-5D-5L). The EQ-5D-5L consists of the EQ-5D descriptive system and the and EQ - Visual Analog Scale (EQ-VAS). The EQ-5D descriptive system consists of 5 different different domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Participants rate their health in each domain which is then combined into a 5-digit score. The EQ-VAS is a measure of patient self-reported health on a vertical scale with endpoints of 100 being 'the best health you can imagine' and zero being 'the worst health you can imagine'. The two scales together represent the participant's self-reported generic QoL.
Kidney disease quality of life. | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 6-months post-intake, 1-, 2-, 3-, 4-, and 5- years post-intake.
  Kidney patients will rate their disease-specific QoL using the Kidney Disease Quality of Life 36-item (KDQOL-36)The KDQOL-36 is scored on a 0-100 scale, with higher scores representing higher QoL. The CLDQ has 5 domains, abdominal symptoms, fatigue, systemic symptoms, activity, emotional function, and worry, and is scored from 1-7, with higher scores indicating higher QoL. The mean of the 5 domains represents overall QoL in liver disease populations.
Liver disease quality of life | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 6-months post-intake, 1-, 2-, 3-, 4-, and 5- years post-intake.
  Liver patients will rate their disease-specific QoL using the Chronic Liver Disease Questionnaire (CLDQ).The CLDQ has 5 domains, abdominal symptoms, fatigue, systemic symptoms, activity, emotional function, and worry, and is scored from 1-7, with higher scores indicating higher QoL. The mean of the 5 domains represents overall QoL in liver disease populations.

SECONDARY OUTCOMES:
Frailty | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 12-weeks post-exercise intervention, 1-year post-exercise intervention
  Frailty as assessed using the Fried Frailty Index and the Liver Frailty Index. Measures of unintentional weight loss, weakness, walking speed, and physical activity during fitness assessments and then calculate a Fried Frailty Index score If present, each criterion is given one point. A total score of equal to or less than one classifies the patient as non-frail, two points is pre-frail, and three or more points is considered frail. For participants who complete the fitness assessments online, a modified version of the Fried Frailty Index, without a measure of weakness, will be used. The Liver Frailty Index will also be used for liver-transplant arm participants. The liver frailty index is a three-variable model which assesses patient frailty based on hand grip strength, balance, and sit-to-stands. Scores range from 1-7, with ≥4.4 is considered frail and a score of 3.2-4.3 is considered pre-frail.
Hand grip strength | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 12-weeks post-exercise intervention, 1-year post-exercise intervention
  Upper body strength will be assessed using a hand grip dynamometer. Participants will complete three trials per side and the highest value in kilograms from each will be taken and added together to get a cumulative value.
Lower extremity flexibility | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 12-weeks post-exercise intervention, 1-year post-exercise intervention
  Chair sit-and-reach test as measured in cm. A reach short of the toes is recorded as a negative value and a reach beyond the toes is recorded as a positive value.
Aerobic Endurance | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 12-weeks post-exercise intervention, 1-year post-exercise intervention
  Participants walk as many laps of a set and measured distance as possible during a six-minute time period.The distance of total laps is added to the final end point for a total distance (metres) walked in six-minutes.
Lower extremity muscular strength | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 12-weeks post-exercise intervention, 1-year post-exercise intervention
  30-second sit-to-stand test. The number of completed sit-to-stands in the 30-second time period is recorded.
Balance | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 12-weeks post-exercise intervention, 1-year post-exercise intervention
  Single-leg stance, double-leg stance, and tandem stance are measured. Each test is a maximum of 20 seconds.
Nutrition | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 6-months post-intake, 1-, 2-, 3-, 4-, and 5- years post-intake.
  Nutrition is measured with the Mini-Eating Assessment Tool (mini-EAT) and the Patient Generated Subjective Global Assessment (PG-SGA). The mini-EAT is a validated brief dietary screener that assesses individuals' consumption of fruits, vegetables, whole grains, refined grains, seafood, legumes/nuts/seeds, low-fat dairy, high-fat dairy, and sweets, with a low-score indicating a poor diet and higher score indicating a healthier diet. The PG-SGA measures nutrition status in hospitalized individuals, classifying individuals as well nourished, moderately or suspected malnourished, or severely malnourished.
Sleep | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 6-months post-intake, 1-, 2-, 3-, 4-, and 5- years post-intake.
  Assessed by Pittsburgh Sleep Quality Index (PSQI). A sum of sleep disturbances over a 1-month period represents an overall sleep quality score.
Mental Health | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 6-months post-intake, 1-, 2-, 3-, 4-, and 5- years post-intake.
  Assessed by Hospital Anxiety and Depression Score. Includes a 7-point anxiety sub-scale and a 7-point depression sub-scale. A score of >8 in a sub-scale indicates anxiety or depression.
Self-efficacy | Study intake, immediately post-exercise intervention, 12-weeks post transplant, 6-months post-intake, 1-, 2-, 3-, 4-, and 5- years post-intake.
  Assessed by a modified exercise barriers self-efficacy scale. 16 items scored on a scale of 1-10 with higher numbers indicating higher self-efficacy to engage in exercise.
Program implementation and evaluation | Baseline to 5-years post exercise intervention
  RE-AIM: reach, effectiveness, adoption, implementation, and maintenance. Reach assessed by enrolment in the TWP, effectiveness measured by primary and secondary outcome individual outcome measures, adoption assessed by number and characteristic of clinics referring to TWP, implementation assessed by fidelity checks , adverse events, time and expertise to deliver intervention, adherence, maintenance assessed by long term self-reported exercise.
Health economic evaluation | Baseline to 5-years post exercise intervention
  Cost-utility of TWP will be assessed by reviews of patient charts to collect health encounters, medication use, emergency room visits, hospital admissions, length of stay, intensive care unit admissions, patient and graft survival over the 5-year follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Mustata, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sim JAP, Perinpanayagam MA, Bahry V, Wytsma-Fisher K, Burak KW, Isaac DL, Mustata S, Culos-Reed SN. An Exercise and Wellness Behavior Change Program for Solid Organ Transplant: A Clinical Research Protocol for the Transplant Wellness Program. Can J Kidney Health Dis. 2024 Oct 21;11:20543581241289196. doi: 10.1177/20543581241289196. eCollection 2024. PMID 39449962